CLINICAL TRIAL: NCT06328621
Title: Lung Cancer Risk Assessment &Amp; Etiology
Brief Title: Lung Cancer Risk Assessment and Etiology
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19594; NCI-2021-05881 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19594 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2024-02-14; First posted 2024-03-25 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (survey, biospecimen, medical record, CT): Participants complete a survey over 40-45 minutes at baseline. Participants' medical records are also reviewed. Participants who have lung cancer but have not undergone treatment and participants not diagnosed with lung cancer (i.e., "unaffected"), undergo collection of blood samples at a scheduled clinical or research blood draw. Participants not diagnosed with lung cancer (i.e. "unaffected"), undergo a low-dose CT scan over 20 minutes.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Electronic Health Record Review; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo low-dose CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Other: Electronic Health Record Review — Review of medical records
Other: Survey Administration — Complete survey

SUMMARY:
This study examines the biological and social determinants that may increase the risk for lung cancer in patients and never-smoking individuals. Biological characteristics of a person can include their genetics and social determinants of a person can include their education, income, and environment, all of which can impact their health. Information collected in this study may help increase early detection of lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the frequency of germline cancer susceptibility mutations in affected and unaffected individuals who have a personal or family history suggestive of high lung cancer risk.

EXPLORATORY OBJECTIVES:

I. To assess the frequency of abnormal radiographic findings in high-risk individuals unaffected with cancer who undergo low-dose computed tomography (CT) screening.

II. Use patient survey and medical record data to explore the associations between social determinants of health, biological risk factors, family history and lung cancer incidence.

III. To determine the sensitivity and specificity of liquid biopsy for detection of lung cancer in a never-smoking population.

OUTLINE:

Participants complete a survey over 40-45 minutes at baseline and undergo collection of blood samples at a scheduled clinical or research blood draw. Participants' medical records are also reviewed. Participants not diagnosed with lung cancer (i.e. "unaffected"), undergo a low-dose computerized tomography (CT) scan over 20 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Have had clinical germline genetic testing and/or have consented or expressed a willingness to consent to the City of Hope (COH) General Research Protocol COH IRB # 07047
* Age >= 18 years
* Willing to have about 30 mL of blood (approximately 2 tablespoons) drawn during the aspiration visit
* Speak English, Spanish, or Mandarin
* Lung cancer patients: meeting at least one of the following criteria:

  * Be a never-smoker with lung cancer (excludes atypical/typical carcinoid and small cell tumors)
  * Be diagnosed with lung cancer =< 50 years of age
  * Have a germline alteration known/suspected to be associated with elevated lung cancer risk
  * Have a strong family history of lung cancer (>= one first, second or third degree relative with never-smoking lung cancer, >= three first, second or third degree relative with lung cancer in one lineage [side of the family], >= one first, second or third degree relative diagnosed with lung cancer under the age of 50. Patients may also be considered eligible if they meet the family history criteria in part and have a truncated family structure [e.g., only one first and one second degree relative with lung cancer in a small family])
* Unaffected patients (i.e., those without a lung cancer diagnosis and other cancer diagnosis for the past 5 years) who are at least 50 years of age or at most age 10 years younger than the first case of lung cancer in the family, meeting at least one of the following criteria:

  * Have a germline alteration known/suspected to be associated with elevated lung cancer risk
  * Have a strong family history of lung cancer (>= one first, second or third degree relative with never-smoking lung cancer, >= three first, second or third degree relative with lung cancer in one lineage [side of the family], >= one first, second or third degree relative diagnosed with lung cancer under the age of 50. Patients may also be considered eligible if they meet the family history criteria in part and have a truncated family structure [e.g., only one first and one second degree relative with lung cancer in a small family])
  * Of East Asian descent with any family history of lung cancer
* Documented informed consent of the participant

Exclusion Criteria:

* Unable to provide informed consent
* Patients who fall under the unaffected cohort criteria but received chest imaging (except chest x-ray) within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Never-smoking patients with and without lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
Frequency of germline alterations | Through study completion, an average of 5 years
  We will explore the relationships between variables, examining correlations (Pearson or Spearman where appropriate). Summarization of data using univariate distributions of the outcomes of interest (presence of lung cancer and molecular phenotypes) and their bivariate distributions with social determinants of health will be carried out. We will examine whether financial hardship, low levels of education, and traffic proximity are associated with presence of lung cancer and molecular phenotypes by using T-tests to compare means and Fisher's exact test to compare proportions. We will also conduct logistic regression modeling to adjust for relevant covariates like race/ethnicity, age, and sex. If appropriate, we will use standard techniques such as sensitivity analyses or multiple imputation to handle missing data.

OTHER OUTCOMES:
Frequency of abnormal radiographic findings | Through study completion, an average of 5 years
  Will assess the frequency of abnormal radiographic findings in high-risk individuals unaffected with cancer who undergo low-dose computed tomography (CT) screening. Will summarize data related to the frequency of abnormal radiographic findings in high-risk individuals who undergo low-dose CT screening.
Associations between molecular phenotypes, social determinants of health, and the presence of lung cancer and related outcomes | Up to study completion
  Identification of associations of social determinants of health and risk factors with lung cancer using lung cancer cases and non cases (survey and medical record data).
Liquid biopsy (LB) test sensitivity | Through study completion, an average of 5 years
  Calculated by comparing the LB results with known cancer status. Results will be reported with their corresponding 95% confidence intervals.
LB test specificity | Through study completion, an average of 5 years
  Calculated by comparing the LB results with known cancer status. Results will be reported with their corresponding 95% confidence intervals.
LB test positive predictive value | Through study completion, an average of 5 years
  Calculated by comparing the LB results with known cancer status. Results will be reported with their corresponding 95% confidence intervals.
LB test negative predictive value | Through study completion, an average of 5 years
  Calculated by comparing the LB results with known cancer status. Results will be reported with their corresponding 95% confidence intervals.
LB test accuracy comparing LB genetic mutations to those found on next generation sequencing (NGS) | Through study completion, an average of 5 years
  LB test sensitivity and specificity, will be calculated by comparing the LB results with known cancer status. In addition to sensitivity and specificity, we will also examine other confusion matrix statistics, such as positive predictive value, negative predictive value, and test accuracy. Results will be reported with their corresponding 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy W Gray, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States